CLINICAL TRIAL: NCT06656962
Title: Renmin Hospital of Wuhan University
Brief Title: The Efficacy and Safety of Treatment with Telitacicept in Antineutrophil Cytoplasmic Antibody-associated Nephritis (AAGN)
Acronym: TEST-T-AAGN
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Huiming Wang, Director, Professor, Renmin Hospital of Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCTAIIRANCA001
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Antineutrophil Cytoplasmic Antibody (ANCA)-associated Nephritis (AAGN)
Keywords: ANCA-associated nephritis; ANCA; Antineutrophil cytoplasmic antibody (ANCA)-associated vasculitis; AAGN
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — telitacicept; Prednisone; Cyclophosphamide; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The Telitacicept treatment group (Experimental)
  Interventions: Drug: Telitacicept 160mg; Drug: Prednisone (and methylprednisolone); Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Telitacicept 160mg — Telitacicept for Injection combined with standard therapy (Prednisone and Cyclophosphamide) for the treatment of ANCA-associated nephritis (AAGN).
  Other Names: Prednisone; Cyclophosphamide
Drug: Prednisone (and methylprednisolone) — Methylprednisone shock therapy (500mg, 3 times), followed by Prednisone (1 mg·kg·d and a pre-determined tapering guideline [PEXIVAS regimen]).
Drug: Cyclophosphamide — Cyclophosphamide, intravenous injection, once every 2 to 3 weeks, 0.75 g/m² each time, the maximum cumulative dose of 8g

SUMMARY:
This study is a prospective, single-arm, open-label exploratory clinical study conducted in subjects with ANCA-associated nephritis (AAGN), aiming to evaluate the efficacy and safety of Telitacicept in the treatment of AAGN.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years, both male and female are included.
2. Clinically diagnosed as granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA) according to the definition of the 2012 Chapel Hill Consensus Conference (CHCC).
3. Positive serological detection of autoantibodies, defined as follows: positive anti-proteinase 3 (PR3-ANCA) or anti-myeloperoxidase (MPO-ANCA) (previous or screening test results).
4. Renal involvement at screening, defined as at least one of the following: (1) At least one renal item in the Birmingham Vasculitis Activity Score (BVAS) version 3.0; (2) According to the pathological classification criteria formulated by the European Vasculitis Society (EUVAS) in 2003, there is active, biopsy-confirmed ANCA-associated nephritis (biopsy must be performed within 1 year before the screening visit or during the screening period); (3) Microscopic examination of urine shows red blood cell casts.
5. Voluntarily participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Life-threatening severe vasculitis (including diffuse alveolar hemorrhage, respiratory failure, intestinal perforation or massive bleeding, cerebral vasculitis, cardiac vasculitis, etc.).
2. Secondary vasculitis (such as systemic lupus erythematosus, Henoch-Schönlein purpura, drugs, tumors, infections, primary immunodeficiency, etc.).
3. Patients with primary kidney diseases (such as IgA nephropathy, membranous nephropathy and anti-glomerular basement membrane nephritis, etc.).
4. Major or uncontrolled diseases unrelated to AAV.
5. Rapidly progressive glomerulonephritis with rapid decline in renal function: estimated glomerular filtration rate (eGFR) ≤ 30 ml/min/1.73m² before the first administration, or already receiving continuous dialysis treatment.
6. Patients with central nervous system diseases (including epilepsy, psychosis, organic brain syndrome, cerebrovascular accident, encephalitis, central nervous system vasculitis).
7. Other multisystem autoimmune diseases including systemic lupus erythematosus, IgA, rheumatoid vasculitis, anti-glomerular basement membrane disease, cryoglobulinemic vasculitis, etc.
8. Active hepatitis or a history of severe liver disease or liver lesions (HBsAg positive, or HBcAb positive and HBV-DNA positive), active pulmonary tuberculosis.
9. Immunodeficiency, uncontrolled severe infection.
10. Abnormal laboratory indicators that need to exclude subjects include but are not limited to the following indicators: total bilirubin ≥ 3 times the upper limit of normal, alanine aminotransferase (ALT) ≥ 3 times the upper limit of normal, aspartate aminotransferase (AST) ≥ 3 times the upper limit of normal, white blood cell (WBC) < 2.5×109/L, hemoglobin (Hb) < 85 g/L, platelet count (PLT) < 50×109/L.
11. Received any of the following treatments within 364 days before day 0: a) B-cell targeted therapy (e.g., rituximab, other anti-CD20 drugs, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], BLyS receptor fusion protein [BR3], TACI-Fc); b) abatacept; c) experimental biological products.
12. Patients who have undergone kidney transplantation or other organ transplantation.
13. Received intravenous immunoglobulin or plasma exchange within 4 weeks before the first administration.
14. Pregnant women, lactating women and men or women with plans for childbearing during the trial.
15. Participated in other new drug clinical trials within 3 months before the first administration.
16. Psychiatric patients with depression or suicidal thoughts.
17. Have a history of major organ (such as heart, lung, kidney, liver) transplantation or hematopoietic stem cell/bone marrow transplantation or plan to receive transplantation.
18. Those with positive test results within 4 weeks before screening suggesting COVID-19 infection, or those with a severe history of COVID-19 requiring hospitalization within 12 months before screening.
19. Those allergic to Telitacicept.
20. Other diseases or conditions that the investigator deems inappropriate for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The complete remission rate of AAGN | 24 weeks
  The complete remission of AAGN is defined as no manifestations of glomerulonephritis (the renal item score of Birmingham vasculitis activity score [BVAS] is 0); the renal item score of BVAS can range from 0 to 58.
The partial remission rate of AAGN | 24 weeks
  The partial remission refers to no active urinary sediment, stable or decreased Scr level, or a reduction of more than 50% in the renal item score of Birmingham vasculitis activity score [BVAS]; the renal item score of BVAS can range from 0 to 58.

SECONDARY OUTCOMES:
The complete remission rate of ANCA | 24 weeks
  The changes of Birmingham vasculitis activity score (BVAS) relative to baseline were calculated, and the proportion of subjects who achieved complete response (BVAS=0); when calculating the total BVAS score, the maximum score for each organ is 12, the total scores can range from 0 to 63.
The partial remission rate of ANCA | 24 weeks
  The partial response (BVAS score decreased by more than 50%) was calculated. The Birmingham Vasculitis Activity Score (BVAS): when calculating the total BVAS score, the maximum score for each organ is 12, the total scores can range from 0 to 63.
Safety and tolerability of patients, occurrence and recurrence of adverse events during the trial | 24 weeks
  This trial specifies that the recording of adverse events shall be recorded as a medical history from the time the subject receives the treatment administration, and from the time of signing the informed consent form until the clinical diagnosis, abnormal signs and symptoms, and examination findings occurring prior to the administration of the induction phase treatment.

OTHER OUTCOMES:
Changes in renal function compared with baseline during follow-up | 48 weeks
  Renal function measures included: 24h urinary total protein (UTP, g/24h), estimated glomerular filtration rate (eGFR, ml/min), serum creatinine (SCr, μmol/L), blood urea nitrogen (BUN, mmol/L), urinary microalbumin/urinary creatinine (UACR, mg/g).
Occurrence of adverse events during follow-up | 48 weeks
  All adverse events were recorded during follow-up, including infection, diarrhea, nausea, rash, prurient, joint pain, dizziness, abnormal liver function, and other drug-related adverse events.
Recurrence of patients during follow-up. | 48 weeks
  Recurrence is defined by a Birmingham vasculitis activity score (BVAS) >15; when calculating the total BVAS score, the maximum score for each organ is 12, the total scores can range from 0 to 63.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided